CLINICAL TRIAL: NCT00767520
Title: A Randomized, Double-Blind, Multi-Center Phase II Trial of Exemestane (AromasinÂ®) Plus Dasatinib Versus Exemestane Plus Placebo in Advanced Estrogen Receptor-Positive Breast Cancer After Disease Progression on a Non-Steroidal Aromatase Inhibitor (NSAI)
Brief Title: Safety and Efficacy of Exemestane Plus Dasatinib Versus Placebo for Advanced ER+ Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA180-261
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Advanced Estrogen Receptor Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Dasatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Exemestane + Dasatinib
- B (Placebo Comparator)
  Interventions: Drug: Exemestane + Placebo

INTERVENTIONS:
Drug: Exemestane + Dasatinib — Tablets, Oral, Exemestane 25 mg + Dasatinib 100 mg, once daily, until disease progression or unacceptable toxicity
  Other Names: Sprycel; BMS-354825
  Arms: A
Drug: Exemestane + Placebo — Tablets, Oral, Exemestane 25 mg + Placebo 100 mg, once daily, until disease progression or unacceptable toxicity
  Arms: B

SUMMARY:
The purpose of this study is to determine whether exemestane plus dasatinib will be well-tolerated and will increase progression-free survival (PFS) in the treatment of advanced estrogen-receptor positive (ER+) breast cancer after disease progression (PD) on a non-steroidal aromatase inhibitor (NSAI).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-documented invasive estrogen receptor positive breast cancer , with tumor tissue from prior surgery available for analysis
* Prior therapy with a non-steroidal aromatase inhibitor
* Recurrent or progressive advanced breast cancer (locally-advanced or metastatic)
* Documented breast cancer with tumor ≤ 28 days prior to study entry
* Women who are NOT of childbearing potential
* Must be able to take oral medication
* Performance Status 0 or 1

Exclusion Criteria:

* Pleural or pericardial effusion or ascites (of any etiology; Grade ≥ 1) within 6 months prior to study entry
* Any chemotherapy, immunotherapy < 6 months before study entry. Any targeted therapy (eg. lapatinib) < 6 months before study entry, unless given in combination with an NSAI
* Any antitumor therapy, including radiotherapy or hormonal therapy, within 15 days prior to study entry
* Prior exposure to exemestane, any Src-family kinase inhibitor including dasatinib, to agents intended to control osteolytic disease other than bisphosphonates, or to any investigational agent for breast cancer
* Concurrent or previous malignant disease requiring chemotherapy or radiation treatment within the prior 3 years
* Significant bleeding disorder, or ongoing or recent clinically-significant gastrointestinal bleeding
* Any serious cardiac condition, including congestive heart failure or myocardial infarction within 6 months, uncontrolled angina, or Class III or IV heart disease as defined by the New York Heart Association, baseline ejection fraction ≤ 40%, diagnosed congenital long QT syndrome, clinically-significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes), QTc interval > 450 msec at baseline (Fridericia correction)
* Hematologic abnormality Grade ≥ 2
* Hypocalcemia of Grade ≥ 1
* Any Chemistry abnormality of Grade ≥ 2 [except Grade 2 indirect bilirubin permitted if diagnosed Gilbert's disease]
* Pregnant Women and Women of Childbearing Potential (WOCBP)
* Extremely lactose intolerant, in the judgment of treating physician (100 mg dasatinib contains 135 mg lactose, posing a problem only if intolerance is severe)
* Receiving any of the following concomitant medications: Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Subjects must discontinue drug use at least 7 days prior to starting dasatinib)
* Potent inhibitors of CYP3A4 isoenzyme
* Prisoners or subjects who are involuntarily incarcerated; or subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (4):
  - Compassionate Cancer Care Medical Group, Inc, Fountain Valley, California
  - Compassionate Cancer Care Medical Group Inc, Riverside, California
  - Pennsylvania Oncology/Hematology Associates, Philadelphia, Pennsylvania
  - The West Clinic, Memphis, Tennessee
- Czechia (2):
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- France (3):
  - Local Institution, Lille
  - Local Institution, Paris
  - Local Institution, Saint-Cloud
- Local Institution, Dublin, Dublin, Ireland
- Poland (3):
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Opole
- Spain (2):
  - Local Institution, Madrid
  - Local Institution, Torrevieja
- Local Institution, Västerås, Sweden
- United Kingdom (3):
  - Local Institution, Chelmsford, Essex
  - Local Institution, London, Greater London
  - Local Institution, Coventry, Warwickshire

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane + Dasatinib: Oral dose of exemestane 25 mg + dasatinib 100 mg, once daily, until disease progression or unacceptable toxicity
- Exemestane + Placebo: Oral dose of exemestane 25 mg + placebo 100 mg, once daily, until disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Started | 79 | 78
Completed | 68 (Completed=Off-treatment; Major reasons: disease progression-50, study drug toxicity-10,AE-3,Death-2) | 61 (Completed=Off-treatment; Major reasons: disease progression-56, study drug toxicity-2,AE-1,Death-1)
Not Completed | 11 | 17
Not completed — Participants still on treatment | 11 | 15
Not completed — Randomized in error and Never treated | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo | Total
Number analyzed (Participants) | 79 | 78 | 157
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline data of 78 participants in the Exemestane + Dasatinib Arm
  Years | 63.2 (12.19) | 60.1 (10.43) | 61.7 (11.41)
Age, Customized [Number; unit: participants]
  < 50 years | 9 | 10 | 19
  >=50 years | 69 | 68 | 137
  Not reported | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 78 | 156
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 68 | 58 | 126
  Asian | 11 | 19 | 30
  Other | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic / Latino | 1 | 0 | 1
  Not Hispanic / Not Latino | 9 | 8 | 17
  Not reported | 69 | 70 | 139
Time from Initial diagnosis to randomization [Mean (Standard Deviation); unit: months] — Baseline data of 76 participants in Exemestane + Placebo Arm
  months | 97.63 (74.866) | 87.09 (64.743) | 92.46 (70.058)
Setting of Non-steroidal Aromatase Inhibitor [Number; unit: participants]
  Adjuvant | 27 | 27 | 54
  Advanced | 52 | 51 | 103
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — The ECOG Performance Status (PS) is used to assess disease severity. A score of 0 is normal activity; 1 is symptoms, but fully ambulatory; 2 is symptomatic, but in bed < 50% of the day; 3 is needs to be in bed > 50% of the day, but not bedridden; 4 is unable to get out of bed; 5 is dead.
  participants
    0=normal activity | 46 | 46 | 92
    1=symptoms, but fully ambulatory | 32 | 30 | 62
    Not reported | 1 | 2 | 3
Symptomatic Bone Disease [Number; unit: participants]
  No | 48 | 46 | 94
  Yes | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Distribution for Exemestane Plus Dasatinib vs Exemestane Plus Placebo
Description: PFS= The time (weeks) from date of randomization to date of progressive disease(PD). PFS for each randomization arm was estimated using the Kaplan-Meier product-limit method. A point estimate and a 95% confidence interval (CI) for the median PFS was computed for each randomization arm using the Brookmeyer & Crowley method. PD=Increase (≥ 20%) in sum of longest diameters from smallest value during study (including baseline).
Time Frame: Prior to study therapy, at 8 week intervals until progression occurs (maximum participant PFS of 71 weeks)
Population: All randomized participants. Participants who died without reporting tumor progression were considered to have progressed on the death date. Participants who neither progressed nor died were censored on the day of their last on-study tumor assessment or the first date of subsequent therapy.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 79 | 78
weeks | 18.1 [15.1 to 24.3] | 16.1 [12.1 to 18.1]
Statistical Analysis 1: Comparison: Exemestane + Dasatinib vs Exemestane + Placebo; Test type: Superiority or Other; p = 0.148, Un-stratified log-rank test; Hazard Ratio (HR) = 0.82

2. Secondary Outcome: Number of Participants With Best Overall Response
Description: Complete response (CR) = Disappearance of all measurable and non-measurable lesions, and no new lesions; Partial response (PR) = Decrease ≥30% from baseline in sum of longest diameters (LD) of all measurable lesions, with neither appearance of new lesions nor unequivocal progression of non-measurable lesions. SD = Disease re-assessment not qualifying as CR, PR or PD(≥20% increase in sum of longest diameters from smallest value).
Time Frame: at 6 months
Population: Response-evaluable participants: All treated participants who had measurable disease at baseline and at least one on-study tumor assessment. Treated participants without on-study tumor assessment due to rapid progression or study drug toxicity were included in the response-evaluable population as non-responders.
Measure: Number; unit: participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 49 | 49
participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 3 | 0
  Stable Disease (SD) | 21 | 14
  Disease Progression | 15 | 23
  Unable to assess | 2 | 1
  Not reported | 8 | 11

3. Secondary Outcome: Percentage of Participants With Clinical Benefit (CB) for Exemestane Plus Dasatinib Arm vs Exemestane Plus Placebo Arm at 6 Months
Description: CB = participants whose best response is CR, PR, or stable disease(SD). CR = Disappearance of all measurable and non-measurable lesions, and no new lesions; PR = Decrease ≥30% from baseline in sum of longest diameters of all measurable lesions, with neither appearance of new lesions nor unequivocal progression of non-measurable lesions. SD = Disease re-assessment not qualifying as CR, PR or PD(≥20% increase in sum of longest diameters from smallest value). Confidence interval computed by Clopper-Pearson method.
Time Frame: at 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 49 | 49
percentage of participants | 30.61 [18.25 to 45.42] | 12.24 [4.63 to 24.77]

4. Secondary Outcome: Percentage of Participants With Response in Exemestane Plus Dasatinib Arm and Exemestane Plus Placebo Arms
Description: Response= Proportion of response-evaluable participants whose best response is CR or PR. Confidence intervals was computed using the Clopper-Pearson method. CR = Disappearance of all measurable and non-measurable lesions, and no new lesions; PR = Decrease ≥30% from baseline in sum of longest diameters of all measurable lesions, with neither appearance of new lesions nor unequivocal progression of non-measurable lesions.
Time Frame: Prior to study therapy, at 8 week intervals until progression occurs (maximum participant response was 39 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 49 | 49
percentage of participants | 6.12 [1.28 to 16.87] | 0 [0 to 0]

5. Secondary Outcome: Participants With Freedom-From-Progression (FFP) at 6 Months
Description: FFP at month 6 is defined for the randomized participants who had the probability of neither progressing nor dying before 6 months.
Time Frame: at 6 months
Reporting Status: Not Posted, anticipated posting 2013-05

6. Secondary Outcome: Time to Response for Exemestane Plus Dasatinib Arm and Exemestane Plus Placebo Arms
Description: Time to response is defined as time from first dose of study therapy until measurement criteria are first met for PR or CR (whichever is recorded first). CR = Disappearance of all measurable and non-measurable lesions, and no new lesions; PR = Decrease ≥30% from baseline in sum of longest diameters of all measurable lesions, with neither appearance of new lesions nor unequivocal progression of non-measurable lesions.
Time Frame: Prior to study therapy, at 8 week intervals until CR or PR. Participants will remain on study (ie, last visit) until disease progression or 30 days after the last dose of study drug, whichever is longer
Reporting Status: Not Posted, anticipated posting 2013-05

7. Secondary Outcome: Duration of Response for Exemestane Plus Dasatinib Arm and Exemestane Plus Placebo Arms
Description: Duration of response is defined as the time from date that measurement criteria are first met for PR or CR until first date of documented PD or death. CR = Disappearance of all measurable and non-measurable lesions, and no new lesions; PR = Decrease ≥30% from baseline in sum of longest diameters of all measurable lesions, with neither appearance of new lesions nor unequivocal progression of non-measurable lesions. PD=Increase (≥ 20%) in sum of longest diameters from smallest value during study (including baseline).
Time Frame: Prior to study therapy, at 8 week intervals. Participants will remain on study (ie, last visit) until disease progression or 30 days after the last dose of study drug, whichever is longer.
Reporting Status: Not Posted, anticipated posting 2013-05

8. Secondary Outcome: Changes in Participant-reported Pain Intensity in Participants With Bone Metastasis
Description: Pain intensity evaluated by administration of the Brief Pain Inventory - Short Form (BPI-sf). The BPI-sf is a psychometrically-validated instrument which measures both pain severity and functional interference caused by pain using an 11-point numerical rating scale. Severity of pain at its "worst", "least" and "on average" in the last 24 hours, and "right now" (ie, at the time the questionnaire is being filled out) is recorded using anchors of "no pain" = "0" and "pain as bad as you can imagine" = "10".
Time Frame: Start of study, at treatment start, after 2, 4, and 8 weeks of therapy and every 8 weeks thereafter, at end-of-treatment. Participants will remain on study (ie, last visit) until disease progression or 30 days after the last dose of study drug.
Reporting Status: Not Posted, anticipated posting 2013-05

9. Secondary Outcome: Changes in Markers of Bone Lysis in Participants With Bone Metastasis
Description: Assay for urinary N-telopeptide was used to evaluate Osteolytic activity.
Time Frame: Screening, Day 1, after week 2, 4, and week 8 and subsequently every 8 weeks, at end-of-treatment. Participants will remain on study (ie, last visit) until disease progression or 30 days after the last dose of study drug.
Reporting Status: Not Posted, anticipated posting 2013-05

10. Secondary Outcome: Number of Participants Who Died, Experienced Serious Adverse Events (SAEs), Adverse Events (AEs) or Discontinuations Due to AEs (as Per National Cancer Institute [NCI] Common Toxicity Criteria for Adverse Events [CTCAE], Version 3.0)
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs were recorded. Grade (GR)1 = mild, GR 2 = moderate, GR 3=severe, GR 4=life threatening, GR 5=death.
Time Frame: From start of study drug therapy up to 30 days after the last dose. Median duration of therapy (on-study time) was 14.29 and 15.29 weeks for dasatinib and placebo groups, respectively.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 79 | 76
participants
  All Deaths | 10 | 2
  All SAEs | 22 | 13
  Drug-related SAEs | 10 | 4
  AEs leading to discontinuation | 20 | 6
  All AEs | 77 | 67
  Drug-related AEs | 70 | 48
  Drug-related Grade 3/4 AEs | 26 | 8
  Drug-related Grade 5 AEs | 0 | 1

11. Secondary Outcome: Number of Participants With Grade 1-4 Hematology Abnormalities (as Per the NCI CTCAE, Version 3.0)
Description: Abnormalities were graded per NCI-CTC, Version 3.0 criteria. Grade (GR)1 = mild, GR 2 = moderate, GR 3 = severe, GR 4 = life threatening. Normal ranges are provided by the Local Laboratory and may vary according to sex and age. Granulocytes, GR 1;<LLN-1.5x 10^9/L, GR 2:<1.5-1.0x10^9/L, GR 3: <1.0 - 0.5x10^9/L, GR, 4: <0.5x10^9 /L; Hemoglobin, GR 1: <LLN-10.0 g/dL, GR 2: <10.0-8.0 g/dL, GR 3: <8.0-6.5 g/dL, GR, 4: <6.5g/dL; Platelets, GR 1: <LLN-75.0x10^9/L, GR 2: <75.0-50.0x10^9/L, GR 3: <50.0-25.0x10^9/L; Leukocytes, GR 1: <LLN-3.0x10^9/L, GR 2: <3.0-2.0x10^9/L, GR 4: <1.0x10^9/L.
Time Frame: Data was collected prior treatment with the study drug, after week 2, 4, and week 8, every 8 weeks thereafter and at the end of the treatment. Median duration (on-study) was 14.29 and 15.29 weeks for dasatinib and placebo groups, respectively.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 79 | 76
participants
  Granulocytes; Grade 1 | 18 | 9
  Granulocytes; Grade 2 | 10 | 1
  Granulocytes; Grade 3 | 2 | 0
  Granulocytes; Grade 4 | 0 | 2
  Granulocytes; Grade Not reported | 2 | 0
  Hemoglobin; Grade 1 | 42 | 21
  Hemoglobin; Grade 2 | 11 | 6
  Hemoglobin; Grade 3 | 1 | 2
  Hemoglobin; Grade 4 | 1 | 2
  Hemoglobin; Grade Not reported | 2 | 0
  Platelet Count; Grade 1 | 10 | 2
  Platelet Count; Grade 2 | 2 | 1
  Platelet Count; Grade 3 | 0 | 1
  Platelet Count; Grade Not reported | 2 | 0
  Leukocytes; Grade 1 | 23 | 12
  Leukocytes; Grade 2 | 7 | 2
  Leukocytes; Grade 4 | 0 | 1
  Leukocytes; Grade Not reported | 2 | 0

12. Secondary Outcome: Number of Participants With Grade 1-4 Serum Chemistry Abnormalities in Alanine Aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase, Bilirubin, Calcium, Creatinine, and Albumin (as Per the NCI CTCAE, Version 3.0)
Description: Grade (GR) 1 = mild, GR 2 = moderate, GR 3 = severe, GR 4 = life threatening). Normal ranges are provided by the Local Laboratory and may vary according to sex and age. Alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase, GR 1: >ULN-2.5 x ULN (upper limit of normal), GR 2: >2.5-5.0 x ULN, GR 3: 5.0-20.0 x ULN; Low calcium, GR 1: <LLN - 8.0 mg/dL, GR 2: <8.0-7.0 mg/dL, GR 4:<6.0 mg/dL; High calcium, GR 1:>ULN - 11.5 mg/dL; bilirubin, GR 1: >ULN-1.5 x ULN,GR 3: >3-10 x ULN; Creatinine, GR1:>ULN-1.5 x ULN, GR2: >1.5-3.0 x ULN; Albumin, GR1:<LLN-3 g/dL,GR2:<3-2 g/dL.
Time Frame: Data was collected prior treatment with the study drug, after week 2, 4, and week 8, every 8 weeks thereafter and at the end of the treatment. Median duration (on-study time) was 14.29 and 15.29 weeks for dasatinib and placebo groups, respectively.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 79 | 76
participants
  Alkaline Phosphatase; Grade 1 | 20 | 15
  Alkaline Phosphatase; Grade 2 | 3 | 10
  Alkaline Phosphatase; Grade 3 | 2 | 0
  Alkaline Phosphatase; Grade Not reported | 2 | 0
  Alanine Aminotransferase; Grade 1 | 38 | 16
  Alanine Aminotransferase; Grade 2 | 4 | 3
  Alanine Aminotransferase; Grade 3 | 0 | 3
  Alanine Aminotransferase; Grade Not reported | 2 | 0
  Aspartate Aminotransferase; Grade 1 | 34 | 18
  Aspartate Aminotransferase; Grade 2 | 7 | 7
  Aspartate Aminotransferase; Grade 3 | 3 | 1
  Aspartate Aminotransferase; Grade Not reported | 2 | 0
  Low Calcium ; Grade 1 | 16 | 6
  Low Calcium ; Grade 2 | 2 | 1
  Low Calcium ; Grade 4 | 1 | 2
  Low Calcium ; Grade Not reported | 2 | 0
  High Calcium ; Grade 1 | 8 | 12
  High Calcium ; Grade Not reported | 2 | 0
  Creatinine; Grade 1 | 13 | 13
  Creatinine; Grade 2 | 3 | 1
  Creatinine; Grade Not reported | 2 | 0
  Bilirubin; Grade 1 | 2 | 6
  Bilirubin; Grade 3 | 0 | 1
  Bilirubin; Grade Not reported | 3 | 0
  Albumin; Grade 1 | 9 | 6
  Albumin; Grade 2 | 6 | 3
  Albumin; Grade Not reported | 2 | 0

13. Primary Outcome: Participants With Disease Progression or Death for Exemestane Plus Dasatinib vs Exemestane Plus Placebo
Description: PD is an increase (≥ 20%) in sum of longest diameters from smallest value during study (including baseline).
Time Frame: Prior to study therapy, at 8 week intervals until progression occurs. Maximum participant PFS of ____ months)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 79 | 78
participants
  Disease Progression | 56 | 59
  Death | 4 | 0
  Censored | 19 | 19

14. Secondary Outcome: Number of Participants With Grade 1-4 Serum Chemistry Abnormalities in Potassium, Magnesium, Sodium, Phosphorous, Uric Acid, and Bicarbonate (as Per the NCI CTCAE, Version 3.0)
Description: Grade (GR)1= mild, GR2= moderate, GR3= severe, GR4= life threatening. Ranges are provided by the local laboratory and may vary according to sex and age. Phosphorous, GR1:<LLN 2.5 mg/dL, GR2:<2.5-2.0 mg/dL, GR3: 1.0-<2.0 mg/dL; Low sodium,GR1:<LLN 130mmol/L, GR3:120-<130 mmol/L; High Magnesium, GR1 >ULN 3.0 mg/dL,GR 3:<0.3 0.8mg/dL; Uric acid, GR1:>ULN 10 mg/dL, GR4:>10 mg/dL; Low potassium, GR1:<LLN 3.0mmol/L,GR3:<3.0 2.5mmol/L; High potassium, GR1:>ULN-5.5 mmol/L, GR2:>5.5-6.0 mmol/L; Bicarbonate, GR1:<LLN-16 mmol/L; GR2:<16 - 11 mmol/L; Hig sodium, GR1:>ULN-150 mmol/L,GR2:>150-155 mmol/L.
Time Frame: as for outcome 12
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Number analyzed (Participants) | 79 | 76
participants
  Low Sodium; Grade 1 | 16 | 10
  Low Sodium; Grade 3 | 1 | 0
  Low Sodium; Grade Not reported | 3 | 0
  Inorganic Phosphorus; Grade 1 | 2 | 1
  Inorganic Phosphorus; Grade 2 | 7 | 8
  Inorganic Phosphorus; Grade 3 | 5 | 1
  Inorganic Phosphorus; Grade Not reported | 3 | 4
  Low Magnesium; Grade 1 | 4 | 6
  Low Magnesium; Grade 3 | 1 | 1
  Low Magnesium; Grade 4 | 0 | 1
  Low Magnesium; Grade Not reported | 7 | 2
  Uric acid; Grade 1 | 16 | 18
  Uric acid; Grade 4 | 2 | 0
  Uric acid; Grade Not reported | 2 | 0
  Low Potassium; Grade 1 | 11 | 4
  Low Potassium; Grade 3 | 1 | 0
  Low Potassium; Grade Not reported | 3 | 0
  High Potassium; Grade 1 | 5 | 6
  High Potassium; Grade 2 | 2 | 0
  High Potassium; Grade Not reported | 3 | 0
  Bicarbonate; Grade 1 | 11 | 8
  Bicarbonate; Grade 2 | 0 | 1
  Bicarbonate; Grade Not reported | 19 | 14
  High Magnesium; Grade 1 | 10 | 5
  High Magnesium; Grade 2 | 2 | 2
  High Magnesium; Grade 3 | 2 | 1
  High Magnesium; Grade Not reported | 7 | 2
  High Sodium; Grade 1 | 2 | 1
  High Sodium; Grade 2 | 1 | 0
  High Sodium; Grade Not reported | 3 | 0

15. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Time Frame: Data was collected prior treatment with the study drug, after week 2, 4, and week 8, every 8 weeks thereafter and at the end of the treatment.
Reporting Status: Not Posted, anticipated posting 2013-05

16. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiograms
Time Frame: as for outcome 15
Reporting Status: Not Posted, anticipated posting 2013-05

ADVERSE EVENTS:
Arm/Group | Exemestane + Dasatinib | Exemestane + Placebo
Serious Adverse Events (participants affected / at risk) | 22/79 | 13/76
Other Adverse Events (participants affected / at risk) | 74/79 | 61/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane + Dasatinib (N=79) | Exemestane + Placebo (N=76)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane + Dasatinib (N=79) | Exemestane + Placebo (N=76)
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10
Decreased appetite (Metabolism and nutrition disorders) | 16 | 8
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Constipation (Gastrointestinal disorders) | 15 | 11
Diarrhoea (Gastrointestinal disorders) | 25 | 7
Oedema peripheral (General disorders) | 7 | 2
Pyrexia (General disorders) | 10 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 20 | 14
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Face oedema (General disorders) | 4 | 0
Hot flush (Vascular disorders) | 4 | 6
Insomnia (Psychiatric disorders) | 8 | 4
Vision blurred (Eye disorders) | 4 | 0
Alanine aminotransferase increased (Investigations) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 5
Nasopharyngitis (Infections and infestations) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 | 1
Rash (Skin and subcutaneous tissue disorders) | 12 | 5
Dizziness (Nervous system disorders) | 6 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0
Fatigue (General disorders) | 18 | 12
Headache (Nervous system disorders) | 21 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Oedema (General disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Bronchitis (Infections and infestations) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 29 | 23
Aspartate aminotransferase increased (Investigations) | 6 | 2
Asthenia (General disorders) | 21 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Influenza like illness (General disorders) | 4 | 0
Palpitations (Cardiac disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.